CLINICAL TRIAL: NCT06109584
Title: Verification of the Correct Insertion of a Supradiaphragmatic Central Venous Catheter by a Single Echocardiographic Plane
Brief Title: Verification of the Correct Insertion of a Central Venous Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Paula Gil Esteller, Principal Investigator, Clinical Professor, Consorci Sanitari de Terrassa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 02-23-270-088
Record Dates: First submitted 2023-10-01; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Catheter Related Complication

STUDY DESIGN:
Intervention Model Description: We propose a prospective diagnostic validity study in which the correct location of the central venous catheter will be verified by ultrasound and then verified by radiography in the same patient, without modifying the usual clinical practice criteria.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVC location with Rx (Active Comparator): After placement of the CVC we will perform the X-ray and subsequent verification of the correct location. Simultaneously, a stopwatch will be started to calculate the time interval until the interpretation of the X-ray by the anesthesiologist.
  Interventions: Device: Insertion of central venous catheter
- CVC location with echocardiography (Active Comparator): Cardiac ultrasound will be performed to visualize the correct position of the CVC tip, and the time until the interpretation of the ultrasound results will also be monitored.
  Interventions: Device: Insertion of central venous catheter

INTERVENTIONS:
Device: Insertion of central venous catheter — Central venous catheter verified by ultrasound and then verified by radiography.

SUMMARY:
The investigators propose a prospective diagnostic validity study in which the correct location of the central venous catheter will be verified by ultrasound and then verified by radiography in the same patient, without modifying the usual clinical practice criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age in whom a decision is made to place a supradiaphragmatic central venous catheter.
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients with devices that may interfere with the ultrasound images.
* Patients with poor ultrasound window
* Patients with superior vena cava syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of malposition of central venous catheter | Through study completion, an average of 1 year
  Incidence of malposition measured by echocardiography and chest radiography in confirming the correct positioning of the tip of the supradiaphragmatic central venous catheter. Moreover, this check can be performed in a shorter time interval.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gil Esteller, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: SAP
Time Frame: In 1 year, for 3 years.
Access Criteria: Anaesthesiologists